CLINICAL TRIAL: NCT04235465
Title: Reliability of the Dynamic Gait Index in Children With Dyslexia
Brief Title: Dynamic Gait Index in Children With Dyslexia
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 02.04.2018 - 112
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Dyslexia; Gait Disorders, Neurologic
Keywords: Dynamic Gait Index; Reliability; Balance; Gait
MeSH Terms: conditions — Dyslexia; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dyslexia Group: 30 patients will be included. Dynamic Gait Index and other assessments will be performed twice with a 7-day interval by two evaluators
  Interventions: Other: Dynamic Gait Index
- Healthy Control Group: 30 healthy children will be included. Dynamic Gait Index will be performed.
  Interventions: Other: Dynamic Gait Index

INTERVENTIONS:
Other: Dynamic Gait Index — The Dynamic Gait Index (DGI) measures functionality and dynamic balance in walking and stair climbing. The DGI consists of 8 items including normal gait on flat ground, gait with speed changes, gait with horizontal head movements, gait with vertical head movements, gait and pivot turn, gait and step over an obstacle, gait around obstacles and steps up and downstairs. The performance on each item is rated on a 4-point scale ranging from 0 (severe disorder) to 3 (independent walking). The total score is 24.

SUMMARY:
The aim of the present study is to investigate reliability in dyslexic children and compare it with healthy peers.

DETAILED DESCRIPTION:
Assessments methods are very important for the detection and treatment of such problems and there is a need for studies that can be applied for the dyslexia group. However fewer attempts have been made to demonstrate the reliability of balance impairments tools in dyslexic children. The DGI is a test that has been used a lot lately because of its minimal requirement for space and equipment, as well as its ability to be used with different patients' groups. The aim of the present study is to investigate reliability in dyslexic children and compare it with healthy peers.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of dyslexia by Child and Adolescent Psychiatry
* Intelligence quotient (IQ)> 85 results of WISC-R
* Age between 8 - 14
* Able to understand the commands given
* Volunteer to study

Exclusion Criteria:

* Having cognitive disorder
* Having neuromuscular disorder
* Having skeletal anomaly
* Having visual or hearing problems

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 30 dyslexia patients, between 8 - 14 years of age, and 30 healthy volunteer peers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The Dynamic Gait Index | Day 0
  The Dynamic Gait Index measures functionality and dynamic balance in walking and stair climbing. The DGI consists of 8 items including normal gait on flat ground, gait with speed changes, gait with horizontal head movements, gait with vertical head movements, gait and pivot turn, gait and step over obstacle, gait around obstacles and steps up and down stairs. The performance on each item is rated on a 4-point scale ranging from 0 (severe disorder) to 3 (independent walking). The total score is 24.
The Dynamic Gait Index | Day 3
  The Dynamic Gait Index measures functionality and dynamic balance in walking and stair climbing. The DGI consists of 8 items including normal gait on flat ground, gait with speed changes, gait with horizontal head movements, gait with vertical head movements, gait and pivot turn, gait and step over obstacle, gait around obstacles and steps up and down stairs. The performance on each item is rated on a 4-point scale ranging from 0 (severe disorder) to 3 (independent walking). The total score is 24.

SECONDARY OUTCOMES:
The Timed Up and Go Test | Day 0
  The Timed Up and Go is a test used to measure mobility and evaluates walking speed, posture control, functional mobility and balance.
Functional Reach Test | Day 0
  Functional Reach Test (FRT) is a static balance test. Measurement is carried out by a tape measure attached to the wall parallel to the floor. The individual was standing parallel to a wall with the feet shoulder wide apart and the shoulders extended at 90 degrees flexion; in this position the third metacarpal head was recorded as the initial position. Then, the patient was asked to reach as forward as (s)he can, without taking a step. Again, the evaluator determined the position of the third metacarpal. The difference in centimeters between the first and second marks determined the FRT value. The FRT was performed three times and average value was taken.

CONTACTS AND LOCATIONS:
Overall Officials: Naime Evrim Karadag-Saygi, Prof, Study Chair — Department of PM&R, Marmara University School of Medicine
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Barela JA, Dias JL, Godoi D, Viana AR, de Freitas PB. Postural control and automaticity in dyslexic children: the relationship between visual information and body sway. Res Dev Disabil. 2011 Sep-Oct;32(5):1814-21. doi: 10.1016/j.ridd.2011.03.011. Epub 2011 Apr 16. PMID 21498044
- [Result] Cattaneo D, Jonsdottir J, Repetti S. Reliability of four scales on balance disorders in persons with multiple sclerosis. Disabil Rehabil. 2007 Dec 30;29(24):1920-5. doi: 10.1080/09638280701191859. Epub 2007 Apr 26. PMID 17852286
- [Result] de Freitas PB, Pedao ST, Barela JA. Visuomotor processing and hand force coordination in dyslexic children during a visually guided manipulation task. Res Dev Disabil. 2014 Oct;35(10):2352-8. doi: 10.1016/j.ridd.2014.06.002. Epub 2014 Jun 22. PMID 24960554
- [Result] Gouleme N, Gerard CL, Bucci MP. The Effect of Training on Postural Control in Dyslexic Children. PLoS One. 2015 Jul 10;10(7):e0130196. doi: 10.1371/journal.pone.0130196. eCollection 2015. PMID 26162071
- [Result] Kapoula Z, Bucci MP. Postural control in dyslexic and non-dyslexic children. J Neurol. 2007 Sep;254(9):1174-83. doi: 10.1007/s00415-006-0460-0. Epub 2007 Aug 3. PMID 17676356